CLINICAL TRIAL: NCT05278793
Title: The Efficacy of Intermittent Versus Daily Oral Iron Supplementation in Anaemic Pregnant Women.
Acronym: FER-IDIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martini Hospital Groningen (Other)
Collaborators: dr. J.M. Munster, gynaecologist, principal investigator (Unknown)
Responsible Party: Principal Investigator, Maryse de Graaf, drs, Martini Hospital Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL77578.000.21; 2021-005393-26 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia; Pregnancy Related
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent (Experimental): This group will receive ferrous fumarate 200mg intermittent three times a week on alternate days.
  Interventions: Drug: Ferrous fumarate
- Daily (Active Comparator): This group will receive ferrous fumarate 200mg once daily.
  Interventions: Drug: Ferrous fumarate

INTERVENTIONS:
Drug: Ferrous fumarate — Ferrous fumarate 200mg oral

SUMMARY:
In this study intermittent dosage of iron supplementation three times a week will be compared to daily dosage in anaemic pregnant women due to iron deficiency.

DETAILED DESCRIPTION:
Background of the study:

Iron deficiency anaemia in pregnancy is common and the standard treatment is iron supplementation once or twice daily. But there is no evidence for the optimal dose of iron supplementation in pregnancy. In non-pregnant women intermittent oral iron supplementation on alternate days is proven to have a similar effect on haemoglobin levels as iron supplementation daily with less side effects. In pregnancy the need and absorption of iron is physiologically higher. Therefore the optimal dose may differ from non-pregnant women.

The adverse effects of iron supplementation, which are mainly gastrointestinal effects, seem to be related to the dose of iron supplementation. These effects often already exist physiologically in pregnancy and may increase with the use of iron supplementation. Therefore, a lower dose would be preferable in pregnancy if the effectiveness is similar.

In this study intermittent dosage of iron supplementation three times a week will be compared to daily dosage in anaemic pregnant women due to iron deficiency. Our hypothesis is that intermittent oral iron supplementation is at least as effective as iron supplementation once daily and will give less adverse effects.

Objective of the study:

To compare the efficacy, side effects and therapy compliance of intermittent (three times a week) versus daily oral iron supplementation for anaemia in pregnancy attributed to iron deficiency.

Study design:

Single-centre, non-inferiority, open-label randomised controlled trial.

Study population:

Pregnant women of 18 years and older with iron deficiency anaemia.

Intervention:

One group will receive ferrous fumarate 200mg intermittent three times a week (for example on Monday, Wednesday and Friday) and one group will receive ferrous fumarate 200mg once daily.

Screening for anaemia during the pregnancy will be done according the local protocol in the first trimester and at a gestational age of 30 weeks. In women at risk for anaemia extra haemoglobin level will be measured at a gestational age of 20 weeks.

When a patient is eligible for the study she will be computer-randomised. Haemoglobin levels will be measured every 6 weeks after the start of the supplementation until the delivery. Side effects and therapy compliance will be evaluated with an interview.

Primary study parameters/outcome of the study:

The main endpoint of the study is the difference in haemoglobin level from baseline to 6 weeks as a continuous variable. A multivariate analysis will be performed with gestational age/trimester at start iron supplementation, the duration of the treatment, use of other supplements, vegetarian diet and the use of proton pump inhibitors or H2 receptor antagonists.

Secondary study parameters/outcome of the study:

The secondary endpoints are haemoglobin level at time of delivery, side effects, therapy compliance, term of delivery, birth weight, parenteral iron ante- or postpartum and blood transfusion postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of 18 years and older
* Iron deficiency anaemia (defined as: Anaemia (haemoglobin lower than cut-off value) AND mean corpuscular volume (MCV) 70-85 fl OR ferritin <30ug/L) OR mean corpuscular volume (MCV) < 70fl / hemoglobinopathy is ruled out.
* Adequate mental health
* Good command of the Dutch language
* No participation in other research with medication
* Informed consent

Exclusion Criteria:

* Start of iron supplementation at pregnancy duration > 37 weeks (because of the limited time to achieve an increase in haemoglobin).
* History of bariatric surgery, inflammatory bowel disease, coeliac disease or Helicobacter pylori infection (because of malabsorption of iron).
* Patients who received blood transfusion or parental iron supplementation during the 3 months prior to screening (because of the effect on the haemoglobin level).
* Patients with significant bleeding, blood donation or surgery during pregnancy (because of the effect on the haemoglobin level).
* Allergy for iron.
* Anaemia of other cause, such as a hemoglobinopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin level | 6 weeks after start treatment
  The main endpoint of the study is the difference in haemoglobin level from baseline to 6 weeks as a continuous variable.

SECONDARY OUTCOMES:
Side effects | 6 weeks after start treatment
  The following treatment related adverse effects will be analysed: headache, dizziness, nausea, vomiting, constipation, diarrhoea. These known side effects of ferrous fumarate will be analysed with a written questionnaire.
Therapy compliance | 6 weeks after start treatment
  Therapy compliance will be analysed with a validated questionnaire (SMAQ).The SMAQ was considered 'positive' when a non-adherent patient was detected, that is, when there was a positive response to any of the qualitative questions (question 1-3), more than two doses missed over the past week, or over 2 days of total non-medication during the past 3 months.
Haemoglobin level at time of delivery | At time of delivery
  When a subject is in labour a haemoglobin level will be measured.
Term of delivery | At delivery
  Gestational age at delivery.
Birth weight | At delivery
  The weight of the neonate.
Parenteral iron ante- or postpartum | From start treatment until 1 week after delivery
  The need for parental iron supplementation when oral supplementation is not sufficient.
Blood transfusion postpartum | Until 1 week after delivery
  The need for a blood transfusion postpartum because of anaemia as binary data (yes / no).

CONTACTS AND LOCATIONS:
Locations (1):
- Martini Hospital Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No